CLINICAL TRIAL: NCT00518505
Title: Long and Short Term Outcomes After Laparoscopic Surgery for Gastroesophageal Reflux Disease
Brief Title: Assessing Outcomes After Surgery for Gastroesophageal Reflux Disorder
Acronym: GERD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Kenneth Luberice, Principal Investigator, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 105238
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Gastroesophageal Reflux Disorder
Keywords: GERD, laparoscopic surgery
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Other): This is a single arm study. All patients will be asked to complete questionnaires and have their medical charts reviewed.
  Interventions: Other: Symptom questionnaire

INTERVENTIONS:
Other: Symptom questionnaire — This questionnaire will assess patient outcomes before and after surgery for gastroesophageal reflux disorder.

SUMMARY:
The purpose of this study is to review pre-operative studies and patient evaluation reports and compare those with the results of the post-operative studies, patient evaluation reports and subjective patients' outcomes following laparoscopic surgery for gastroesophageal reflux disorder. This will allow us to evaluate how patients have benefited from the procedure.

DETAILED DESCRIPTION:
This study will include all patients who have laparoscopic surgery for gastroesophageal reflux disorder. Patients who participate will be asked to answer questionnaires regarding symptoms of reflux before and after surgery. In addition medical charts will be reviewed for relevant data.

ELIGIBILITY:
Inclusion Criteria:

* patients must have GERD and must plan to have laparoscopic surgery for GERD.
* patients must be at least 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2006-12; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The objective of this study is to review pre-operative studies and evaluation reports and compare those with post-operative studies and evaluation reports to evaluate outcome following laparoscopic surgery for GERD. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Rosemurgy, M.D., Study Director — University of South Florida
Locations (1):
- Tampa General Hospital/University of South Florida, Tampa, Florida, United States